CLINICAL TRIAL: NCT03117816
Title: Efficacy and Safety of Pegylated Proline Interferon Alpha 2b (AOP2014) in Maintaining Deep Molecular Remissions in Patients With Chronic Myeloid Leukemia (CML) Who Discontinue ABL-Kinase Inhibitor Therapy - a Randomized Phase III, Multicenter Trial With Post-study Follow-up
Brief Title: ENDURE - Efficacy and Safety of AOP2014 With CML Patients in Remission
Acronym: ENDURE-CML-IX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Principal Investigator, Kerstin Balthasar, KKS Marburg Sponsor representative, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KKS-227; 2016-001030-94 (EudraCT Number)
Record Dates: First submitted 2017-03-08; First posted 2017-04-18 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Chronic Myeloid Leukemia in Remission
Keywords: deep molecular remission of MR4 or better

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A randomized, open-label assessor blinded, multi-center, controlled phase III trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- investigational arm A (Experimental): There will be an overlapping treatment with AOP2014 and TKI for one month. After one month, the TKI therapy will be stopped and patient will receive only AOP2014 treatment for the next 14 months.
  Interventions: Drug: AOP2014 / Pegylated-Proline-interferon alpha-2b
- surveillance arm B (Other): This is an open-label study with a "surveillance" group as comparator arm. Similar as in the arm A, patient will discontinue TKI therapy one month after randomization. From then on patient will receive no further CML treatment.
  Interventions: Other: Surveillance

INTERVENTIONS:
Drug: AOP2014 / Pegylated-Proline-interferon alpha-2b — AOP2014 as pre-filled auto-injection pen for subcutaneous injection, containing 250 µg AOP2014 / 0.5 ml. The solution also contains inactive ingredients (sodium chloride, polysorbate 80, benzyl alcohol, sodium acetate, and acetic acid). The solution is colorless to light yellow.
  Arms: investigational arm A
Other: Surveillance — For patients randomized into this treatment arm stopp their standard treatment and will just be under observation.
  Arms: surveillance arm B

SUMMARY:
A randomized, open-label assessor blinded, multi-center, controlled phase III Trial to evaluate the efficacy of AOP2014 administered bi-weekly subcutaneously (s.c.) in preventing molecular relapse (loss of MMR) in CML patients, who discontinue ABL tyrosine kinase inhibitor therapy (TKI) in deep molecular remission of MR4 or better (MR4.5, or MR5).

DETAILED DESCRIPTION:
Four hypotheses are tested in hierarchical order. To avoid inflation of type 1 error (false rejection of a null hypothesis), further confirmatory testing has to be stopped as soon as a null hypothesis could not be rejected.

All four hypotheses are tested at significance level 0.05. Null hypothesis 1 is the primary endpoint and investigates molecular relapse-free survival as a time-to-event variable; the two arms are compared with the log-rank test. Null hypotheses 2, 3, and 4 deal with probabilities of molecular relapse-free survival 7, 13, and 25 months after randomization, respectively; arms A and B are compared with the uncorrected chi-square test.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form.
2. Capability and willingness to comply with study procedures and ability to self-administration of the study drug.
3. Male or female aged ≥ 18 years.
4. At least three years of TKI therapy.
5. BCR-ABL-positive, chronic phase CML patients with a transcript level according to the international scale (IS) of at least MR4, or better (MR4.5, MR5). MR4 is defined as (i) detectable disease ≤0.01% BCR-ABL IS or (ii) undetectable disease in cDNA with ≥10,000 ABL or ≥24,000 GUS transcripts for at least one year. There have to be at least three consecutive PCR-results with MR4 or better within the last year (+ months) before study entry. The latest of these PCRs must be a confirmatory MR4 measurement prior to randomization by the EUTOS-certified Study Reference Laboratories for PCR (BCR-ABL mRNA). No PCR-results in the last year before randomisation can be worse than MR4. If the last PCR was not done within two months from baseline (day 0) in an EUTOS-certified study Reference Laboratory; the PCR sample must be sent to an EUTOS-certified study Reference Laboratory at screening.
6. Patients who had failed to discontinue TKI in a prior discontinuation attempt are eligible for this protocol, if they fulfil criterion 5 after retreatment with TKI. A prior TKI discontinuation failure must be specifically indicated at inclusion and documented.
7. Adequate organ function:

   especially total bilirubin, lactate dehydrogenase [LDH], aspartate aminotransferase [AST], alanine aminotransferase [ALT] and coagulation parameters ≤ 2 × upper limit of normal (ULN)
8. Adequate hematological parameters:

   platelet count ≥ 100 × 1000000000/L; white blood cell count ≥ 2.5 × 1000000000/L; lymphocytes ≥ 1.0 × 1000000000/L; hemoglobin ≥ 9.0 g/dL or 5.59 mmol/L.
9. Female patients with reproductive potential must agree to maintain highly effective methods of contraception by practicing abstinence or by using at least two methods of birth control from the date of consent through the end of the study. If abstinence could not be practiced, a combination of hormonal contraceptive (oral, injectable, or implants) and a barrier method (condom, diaphragm with a vaginal spermicidal agent) has to be used. Male patients must agree to use condoms during study participation.
10. Negative serum pregnancy test in women of childbearing potential.
11. Date of diagnosis of CML confirmed by laboratory PCR must be known.

Exclusion Criteria:

1. Rare variants of BCR-ABL not quantifiable by RT-PCR according to the international scale (IS).
2. Current or previous autoimmune diseases requiring treatment.
3. Immunosuppressive treatment of any kind; transplant recipients
4. Prior allogeneic stem cell transplantation.
5. Prior pegylated IFN therapy. Prior low dose conventional IFN treatment with ≤ 3 x 3 Mio I.E. / week for less than 1 year is acceptable.
6. History of TKI resistance within the last 4 years of TKI therapy.
7. History of accelerated phase or blast crisis.
8. Hypersensitivity/allergy to the active substance or excipients of the formulation.
9. Severe hepatic dysfunction or decompensated cirrhosis.
10. End stage renal disease (GFR <15 ml/min)
11. Thyroid disease that cannot be controlled by conventional therapy.
12. Uncontrolled diabetes mellitus
13. Epilepsy or other disorders of the central nervous system.
14. Severe cardiac disease history including unstable or uncontrolled cardiac disease in the previous 6 months.
15. Uncontrolled hypertension
16. Any history of retinopathy e.g. retinal detachment, degeneration or thromboembolic events.
17. Clinically significant concomitant diseases or conditions, which, in the opinion of the investigator, would lead to an unacceptable risk for the patient to participate in the study (please refer also to the actual Investigator Brochure).
18. Other malignancy, except adequately treated superficial bladder cancer, basal or squamous cell carcinoma of the skin, or other cancer(s) for which the patient has been disease free for more than 3 years.
19. Active or uncontrolled infections at the time of randomization.
20. Pregnant and/or nursing women.
21. Use of antibiotic therapy within the last 2 weeks prior to randomization
22. Concurrent use of molecular targeted therapy.
23. Tested HIV sero-positivity or tested active hepatitis B or C infection.
24. Participation in another clinical study with other investigational drugs within 14 days prior to randomization.
25. Vaccination within 1 month prior to randomization.
26. Any medical, mental, psychological or psychiatric condition (particularly severe depression, suicidal ideation or suicide attempt) that in the opinion of the investigator would not permit the patient to complete the study or comply to study procedures.
27. Drug and/or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
mRFS | Randomization until time of relapse
  The primary efficacy endpoint is molecular relapse free survival (mRFS). Relapse is defined as loss of major molecular remission, MMR, which is any increase of the BCR-ABL ratio to > 0.1% according to the international scale (IS). Time to relapse is defined as the time from randomization to relapse the BCR-ABL ratio to > 0.1% according to the international scale (IS). Time to relapse is defined as the time from randomization to relapse.

SECONDARY OUTCOMES:
mRFS 7 | 7 months after randomization
  The primary efficacy endpoint is molecular relapse free survival, RFS 7 months after
mRFS 13 | 13 months after randomization
  The relapse free survival, RFS 13 months after randomization
mRFS 25 | 25 months after randomization
  The relapse free survival, RFS 25 months after randomization
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | Day 0 - Month 15 (Arm B) or Month 16 (additional safety visit one month after last application for Arm A)
  Adverse events, serious adverse events (AEs, SAEs)• Safety, tolerability and toxicity based on incidences of adverse events, serious adverse events
Quality of life measured by EORTC QLQ-C30 | Day 0 - Month 25
  The QoL assessment in this study is planned to gain information on the QoL of CML patients under stopping conditions. The data will be compared between the treatment groups and to QoL of normal population.
Quality of life measured by EORTC-QLQ-CML24 | Day 0 - Month 25
  The QoL assessment in this study is planned to gain information on the QoL of CML patients under stopping conditions. The data will be compared between the treatment groups and to QoL of normal population. Furthermore, results of the CML24 module should be shared with the EORTC group to complete the validation of this questionnaire
OS (overall survival) | Day 0 - Month 25 (plus annual post study follow up Months 36,48,60)
  Overall survival (OS), defined as the time between the date of randomization and the date of death from any cause.
Kinetics of BCR-ABL transcript level over time after TKI stop | Day 0 - Month 25 (plus annual post study follow up Months 36,48,60)
  Kinetics of BCR-ABL transcript level over time after TKI stop
For Germany: Detection of blood parameters 95 CD86+pDC as mRFS predictor | Day 0 - Month 25 (plus annual post study follow up Months 36,48,60)
  For Germany: To explore the value of 95 CD86+pDC / 105 lymphocytes at baseline in predicting risk of molecular relapse (loss of MMR)
For Germany: Explore immunological and genetic biomarkers and identify predictors | Day 0 - Month 25 (plus annual post study follow up Months 36,48,60)
  For Germany: Explore immunological and genetic biomarkers to study biology of TFR, and identify predictors IFN response (e.g. mRNA sequencing of whole blood or leukocyte subpopulations, PD-L1-, PD1-, CD62L- measurements by FACS on peripheral blood subsets, T-cell activation and exhaustion marker measurements, PR1-CTL assessment and cytokines). Evaluation of cytokines/chemokines (i.e., IL-6, IFN-α, IL 10, and others).
For Germany: Evaluation of cytokines/chemokines | Day 0 - Month 25 (plus annual post study follow up Months 36,48,60)
  For Germany: Evaluation of cytokines/chemokines (i.e., IL-6, IFN-α, IL 10, and others)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Burchert, Prof. Dr., Study Director — Philipps University Marburg; Franck E Nicoloni, MD, PhD, Principal Investigator — Centre Léon Bérard, Lyon
Locations (26):
- France (3):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - CHRU de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (23):
  - 03 Universitätsklinikum Aachen, Hämatologie/Onkologie, Aachen
  - 18 Studienzentrum Aschaffenburg, Aschaffenburg
  - 06 Universitätsmedizin Berlin Charite- Campus Virchow Klinikum, Klinik für Hämatologie und Onkologie, Berlin
  - 19 Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik III, Bonn
  - 16 Klinikum Bremen Mitte, Medizinische Klinik I, Bremen
  - 22 BAG / Onkologische Gemeinschaftspraxis, Dresden
  - 05 Universitätsklinikum Düsseldorf, Klinik für Hämatologie, Onkologie und Klinische Immunologie, Düsseldorf
  - 07 Universitätsklinikum Erlangen, Medizinische Klinik 5, Erlangen
  - 20 Universitätsklinikum Essen, Klinik für Hämatologie, Essen
  - 17 Klinikum der Goethe Universität, Medizinische Klinik II, Frankfurt A. Main
  - 21 Universitätsklinikum Hamburg Eppendorf, Klinik für Onkologie, Hämatologie und KMT, Hamburg
  - 23 Evangelische Krankenhaus Hamm gGmbH, Klinik für Hämatologie, Onkologie und Palliativmedizin, Hamm
  - 02 Universitätsklinikum Jena, linik für Innere Medizin II Abt. für Hämatologie und Internistische Onkologie, Jena
  - 24 Institut für Versorgungsforschung in der Onkologie GbR, Koblenz
  - 13 Universitätsklinikum Leipzig, Abteilung für Hämatologie u. Internistische Onkologie, Leipzig
  - 14 Johannes-Gutenberg-Universität III. Medizinische Klinik, Mainz
  - 04 Universitätsmedizin Mannheim, III. Medizinische Klinik, Mannheim
  - 01 Universitätsklinikum Gießen und Marburg GmbH, Standort Marburg, Klinik für Hämatologie, Onkologie und Immunologie, Marburg
  - 10 Technische Universität München (TUM) Klinikum rechts der Isar, III. Medizinische Klinik und Poliklinik, Munich
  - 08 Universitätsklinikum Münster, Medizinische Klinik, Innere Medizin A, Münster
  - 09 Universitätsklinikum Tübingen, Medizinische Klinik, Tübingen
  - 12 Universitätsklinikum Ulm, Klinik für Innere Medizin III, Ulm
  - 15 Universitätsklinikum Würzburg, Zentrum für Innere Medizin, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben-Neriah Y, Daley GQ, Mes-Masson AM, Witte ON, Baltimore D. The chronic myelogenous leukemia-specific P210 protein is the product of the bcr/abl hybrid gene. Science. 1986 Jul 11;233(4760):212-4. doi: 10.1126/science.3460176.
- [Background] Daley GQ, Van Etten RA, Baltimore D. Induction of chronic myelogenous leukemia in mice by the P210bcr/abl gene of the Philadelphia chromosome. Science. 1990 Feb 16;247(4944):824-30. doi: 10.1126/science.2406902.
- [Background] Perrotti D, Jamieson C, Goldman J, Skorski T. Chronic myeloid leukemia: mechanisms of blastic transformation. J Clin Invest. 2010 Jul;120(7):2254-64. doi: 10.1172/JCI41246. Epub 2010 Jul 1. PMID 20592475
- [Background] Saussele S, Lauseker M, Gratwohl A, Beelen DW, Bunjes D, Schwerdtfeger R, Kolb HJ, Ho AD, Falge C, Holler E, Schlimok G, Zander AR, Arnold R, Kanz L, Dengler R, Haferlach C, Schlegelberger B, Pfirrmann M, Muller MC, Schnittger S, Leitner A, Pletsch N, Hochhaus A, Hasford J, Hehlmann R; German CML Study Group. Allogeneic hematopoietic stem cell transplantation (allo SCT) for chronic myeloid leukemia in the imatinib era: evaluation of its impact within a subgroup of the randomized German CML Study IV. Blood. 2010 Mar 11;115(10):1880-5. doi: 10.1182/blood-2009-08-237115. Epub 2009 Nov 18. PMID 19965667
- [Background] Hochhaus A, O'Brien SG, Guilhot F, Druker BJ, Branford S, Foroni L, Goldman JM, Muller MC, Radich JP, Rudoltz M, Mone M, Gathmann I, Hughes TP, Larson RA; IRIS Investigators. Six-year follow-up of patients receiving imatinib for the first-line treatment of chronic myeloid leukemia. Leukemia. 2009 Jun;23(6):1054-61. doi: 10.1038/leu.2009.38. Epub 2009 Mar 12. PMID 19282833
- [Background] Larson RA, Hochhaus A, Hughes TP, Clark RE, Etienne G, Kim DW, Flinn IW, Kurokawa M, Moiraghi B, Yu R, Blakesley RE, Gallagher NJ, Saglio G, Kantarjian HM. Nilotinib vs imatinib in patients with newly diagnosed Philadelphia chromosome-positive chronic myeloid leukemia in chronic phase: ENESTnd 3-year follow-up. Leukemia. 2012 Oct;26(10):2197-203. doi: 10.1038/leu.2012.134. Epub 2012 May 18. PMID 22699418
- [Background] Jabbour E, Kantarjian HM, Saglio G, Steegmann JL, Shah NP, Boque C, Chuah C, Pavlovsky C, Mayer J, Cortes J, Baccarani M, Kim DW, Bradley-Garelik MB, Mohamed H, Wildgust M, Hochhaus A. Early response with dasatinib or imatinib in chronic myeloid leukemia: 3-year follow-up from a randomized phase 3 trial (DASISION). Blood. 2014 Jan 23;123(4):494-500. doi: 10.1182/blood-2013-06-511592. Epub 2013 Dec 5. PMID 24311723
- [Background] Baccarani M, Deininger MW, Rosti G, Hochhaus A, Soverini S, Apperley JF, Cervantes F, Clark RE, Cortes JE, Guilhot F, Hjorth-Hansen H, Hughes TP, Kantarjian HM, Kim DW, Larson RA, Lipton JH, Mahon FX, Martinelli G, Mayer J, Muller MC, Niederwieser D, Pane F, Radich JP, Rousselot P, Saglio G, Saussele S, Schiffer C, Silver R, Simonsson B, Steegmann JL, Goldman JM, Hehlmann R. European LeukemiaNet recommendations for the management of chronic myeloid leukemia: 2013. Blood. 2013 Aug 8;122(6):872-84. doi: 10.1182/blood-2013-05-501569. Epub 2013 Jun 26. PMID 23803709
- [Background] Cross NC, White HE, Muller MC, Saglio G, Hochhaus A. Standardized definitions of molecular response in chronic myeloid leukemia. Leukemia. 2012 Oct;26(10):2172-5. doi: 10.1038/leu.2012.104. Epub 2012 Apr 16. PMID 22504141
- [Background] Muller MC, Cross NC, Erben P, Schenk T, Hanfstein B, Ernst T, Hehlmann R, Branford S, Saglio G, Hochhaus A. Harmonization of molecular monitoring of CML therapy in Europe. Leukemia. 2009 Nov;23(11):1957-63. doi: 10.1038/leu.2009.168. Epub 2009 Aug 27. PMID 19710700
- [Background] Hehlmann R, Muller MC, Lauseker M, Hanfstein B, Fabarius A, Schreiber A, Proetel U, Pletsch N, Pfirrmann M, Haferlach C, Schnittger S, Einsele H, Dengler J, Falge C, Kanz L, Neubauer A, Kneba M, Stegelmann F, Pfreundschuh M, Waller CF, Spiekermann K, Baerlocher GM, Ehninger G, Heim D, Heimpel H, Nerl C, Krause SW, Hossfeld DK, Kolb HJ, Hasford J, Saussele S, Hochhaus A. Deep molecular response is reached by the majority of patients treated with imatinib, predicts survival, and is achieved more quickly by optimized high-dose imatinib: results from the randomized CML-study IV. J Clin Oncol. 2014 Feb 10;32(5):415-23. doi: 10.1200/JCO.2013.49.9020. Epub 2013 Dec 2. PMID 24297946
- [Background] Graham SM, Jorgensen HG, Allan E, Pearson C, Alcorn MJ, Richmond L, Holyoake TL. Primitive, quiescent, Philadelphia-positive stem cells from patients with chronic myeloid leukemia are insensitive to STI571 in vitro. Blood. 2002 Jan 1;99(1):319-25. doi: 10.1182/blood.v99.1.319. PMID 11756187
- [Background] Corbin AS, Agarwal A, Loriaux M, Cortes J, Deininger MW, Druker BJ. Human chronic myeloid leukemia stem cells are insensitive to imatinib despite inhibition of BCR-ABL activity. J Clin Invest. 2011 Jan;121(1):396-409. doi: 10.1172/JCI35721. Epub 2010 Dec 13. PMID 21157039
- [Background] Cortes J, O'Brien S, Kantarjian H. Discontinuation of imatinib therapy after achieving a molecular response. Blood. 2004 Oct 1;104(7):2204-5. doi: 10.1182/blood-2004-04-1335. No abstract available. PMID 15377577
- [Background] Rousselot P, Huguet F, Rea D, Legros L, Cayuela JM, Maarek O, Blanchet O, Marit G, Gluckman E, Reiffers J, Gardembas M, Mahon FX. Imatinib mesylate discontinuation in patients with chronic myelogenous leukemia in complete molecular remission for more than 2 years. Blood. 2007 Jan 1;109(1):58-60. doi: 10.1182/blood-2006-03-011239. Epub 2006 Sep 14. PMID 16973963
- [Background] Mahon FX, Rea D, Guilhot J, Guilhot F, Huguet F, Nicolini F, Legros L, Charbonnier A, Guerci A, Varet B, Etienne G, Reiffers J, Rousselot P; Intergroupe Francais des Leucemies Myeloides Chroniques. Discontinuation of imatinib in patients with chronic myeloid leukaemia who have maintained complete molecular remission for at least 2 years: the prospective, multicentre Stop Imatinib (STIM) trial. Lancet Oncol. 2010 Nov;11(11):1029-35. doi: 10.1016/S1470-2045(10)70233-3. Epub 2010 Oct 19. PMID 20965785
- [Background] Ross DM, Branford S, Seymour JF, Schwarer AP, Arthur C, Yeung DT, Dang P, Goyne JM, Slader C, Filshie RJ, Mills AK, Melo JV, White DL, Grigg AP, Hughes TP. Safety and efficacy of imatinib cessation for CML patients with stable undetectable minimal residual disease: results from the TWISTER study. Blood. 2013 Jul 25;122(4):515-22. doi: 10.1182/blood-2013-02-483750. Epub 2013 May 23. PMID 23704092
- [Background] Rousselot P, Charbonnier A, Cony-Makhoul P, Agape P, Nicolini FE, Varet B, Gardembas M, Etienne G, Rea D, Roy L, Escoffre-Barbe M, Guerci-Bresler A, Tulliez M, Prost S, Spentchian M, Cayuela JM, Reiffers J, Chomel JC, Turhan A, Guilhot J, Guilhot F, Mahon FX. Loss of major molecular response as a trigger for restarting tyrosine kinase inhibitor therapy in patients with chronic-phase chronic myelogenous leukemia who have stopped imatinib after durable undetectable disease. J Clin Oncol. 2014 Feb 10;32(5):424-30. doi: 10.1200/JCO.2012.48.5797. Epub 2013 Dec 9. PMID 24323036
- [Background] Branford S, Yeung DT, Ross DM, Prime JA, Field CR, Altamura HK, Yeoman AL, Georgievski J, Jamison BA, Phillis S, Sullivan B, Briggs NE, Hertzberg M, Seymour JF, Reynolds J, Hughes TP. Early molecular response and female sex strongly predict stable undetectable BCR-ABL1, the criteria for imatinib discontinuation in patients with CML. Blood. 2013 May 9;121(19):3818-24. doi: 10.1182/blood-2012-10-462291. Epub 2013 Mar 20. PMID 23515925
- [Background] Talpaz M, Kantarjian HM, McCredie KB, Keating MJ, Trujillo J, Gutterman J. Clinical investigation of human alpha interferon in chronic myelogenous leukemia. Blood. 1987 May;69(5):1280-8. PMID 3471281
- [Background] Talpaz M, Kantarjian HM, McCredie K, Trujillo JM, Keating MJ, Gutterman JU. Hematologic remission and cytogenetic improvement induced by recombinant human interferon alpha A in chronic myelogenous leukemia. N Engl J Med. 1986 Apr 24;314(17):1065-9. doi: 10.1056/NEJM198604243141701. PMID 3457264
- [Background] Hehlmann R, Heimpel H, Hasford J, Kolb HJ, Pralle H, Hossfeld DK, Queisser W, Loffler H, Hochhaus A, Heinze B, et al. Randomized comparison of interferon-alpha with busulfan and hydroxyurea in chronic myelogenous leukemia. The German CML Study Group. Blood. 1994 Dec 15;84(12):4064-77. PMID 7994025
- [Background] Guilhot F, Chastang C, Michallet M, Guerci A, Harousseau JL, Maloisel F, Bouabdallah R, Guyotat D, Cheron N, Nicolini F, Abgrall JF, Tanzer J. Interferon alfa-2b combined with cytarabine versus interferon alone in chronic myelogenous leukemia. French Chronic Myeloid Leukemia Study Group. N Engl J Med. 1997 Jul 24;337(4):223-9. doi: 10.1056/NEJM199707243370402. PMID 9227927
- [Background] Hughes TP, Kaeda J, Branford S, Rudzki Z, Hochhaus A, Hensley ML, Gathmann I, Bolton AE, van Hoomissen IC, Goldman JM, Radich JP; International Randomised Study of Interferon versus STI571 (IRIS) Study Group. Frequency of major molecular responses to imatinib or interferon alfa plus cytarabine in newly diagnosed chronic myeloid leukemia. N Engl J Med. 2003 Oct 9;349(15):1423-32. doi: 10.1056/NEJMoa030513. PMID 14534335
- [Background] Hochhaus A, Reiter A, Saussele S, Reichert A, Emig M, Kaeda J, Schultheis B, Berger U, Shepherd PC, Allan NC, Hehlmann R, Goldman JM, Cross NC. Molecular heterogeneity in complete cytogenetic responders after interferon-alpha therapy for chronic myelogenous leukemia: low levels of minimal residual disease are associated with continuing remission. German CML Study Group and the UK MRC CML Study Group. Blood. 2000 Jan 1;95(1):62-6. PMID 10607685
- [Background] Bonifazi F, de Vivo A, Rosti G, Guilhot F, Guilhot J, Trabacchi E, Hehlmann R, Hochhaus A, Shepherd PC, Steegmann JL, Kluin-Nelemans HC, Thaler J, Simonsson B, Louwagie A, Reiffers J, Mahon FX, Montefusco E, Alimena G, Hasford J, Richards S, Saglio G, Testoni N, Martinelli G, Tura S, Baccarani M; Europena Study Group on Interferon in Chronic Myeloid Leukemia; Italian Cooperative Study Group on CML; France Intergroup of CML; German CML Study Group; UK Medical Research Council Working Party on CML; Spanish CML Study Group; Australian CML Study Group; Swedish CML Study Group. Chronic myeloid leukemia and interferon-alpha: a study of complete cytogenetic responders. Blood. 2001 Nov 15;98(10):3074-81. doi: 10.1182/blood.v98.10.3074. PMID 11698293
- [Background] Mahon FX, Delbrel X, Cony-Makhoul P, Faberes C, Boiron JM, Barthe C, Bilhou-Nabera C, Pigneux A, Marit G, Reiffers J. Follow-up of complete cytogenetic remission in patients with chronic myeloid leukemia after cessation of interferon alfa. J Clin Oncol. 2002 Jan 1;20(1):214-20. doi: 10.1200/JCO.2002.20.1.214. PMID 11773172
- [Background] Mauro MJ, Druker BJ, Maziarz RT. Divergent clinical outcome in two CML patients who discontinued imatinib therapy after achieving a molecular remission. Leuk Res. 2004 May;28 Suppl 1:S71-3. doi: 10.1016/j.leukres.2003.10.017. PMID 15036945
- [Background] Merante S, Orlandi E, Bernasconi P, Calatroni S, Boni M, Lazzarino M. Outcome of four patients with chronic myeloid leukemia after imatinib mesylate discontinuation. Haematologica. 2005 Jul;90(7):979-81. PMID 15996937
- [Background] Burchert A, Wolfl S, Schmidt M, Brendel C, Denecke B, Cai D, Odyvanova L, Lahaye T, Muller MC, Berg T, Gschaidmeier H, Wittig B, Hehlmann R, Hochhaus A, Neubauer A. Interferon-alpha, but not the ABL-kinase inhibitor imatinib (STI571), induces expression of myeloblastin and a specific T-cell response in chronic myeloid leukemia. Blood. 2003 Jan 1;101(1):259-64. doi: 10.1182/blood-2002-02-0659. Epub 2002 Jun 28. PMID 12393722
- [Background] Molldrem JJ, Lee PP, Wang C, Felio K, Kantarjian HM, Champlin RE, Davis MM. Evidence that specific T lymphocytes may participate in the elimination of chronic myelogenous leukemia. Nat Med. 2000 Sep;6(9):1018-23. doi: 10.1038/79526. PMID 10973322
- [Background] Molldrem JJ, Lee PP, Kant S, Wieder E, Jiang W, Lu S, Wang C, Davis MM. Chronic myelogenous leukemia shapes host immunity by selective deletion of high-avidity leukemia-specific T cells. J Clin Invest. 2003 Mar;111(5):639-47. doi: 10.1172/JCI16398. PMID 12618518
- [Background] Kreutzman A, Rohon P, Faber E, Indrak K, Juvonen V, Kairisto V, Voglova J, Sinisalo M, Flochova E, Vakkila J, Arstila P, Porkka K, Mustjoki S. Chronic myeloid leukemia patients in prolonged remission following interferon-alpha monotherapy have distinct cytokine and oligoclonal lymphocyte profile. PLoS One. 2011;6(8):e23022. doi: 10.1371/journal.pone.0023022. Epub 2011 Aug 9. PMID 21857985
- [Background] Baccarani M, Martinelli G, Rosti G, Trabacchi E, Testoni N, Bassi S, Amabile M, Soverini S, Castagnetti F, Cilloni D, Izzo B, de Vivo A, Messa E, Bonifazi F, Poerio A, Luatti S, Giugliano E, Alberti D, Fincato G, Russo D, Pane F, Saglio G; GIMEMA Working Party on Chronic Myeloid Leukemia. Imatinib and pegylated human recombinant interferon-alpha2b in early chronic-phase chronic myeloid leukemia. Blood. 2004 Dec 15;104(13):4245-51. doi: 10.1182/blood-2004-03-0826. Epub 2004 Aug 19. PMID 15319292
- [Background] Preudhomme C, Guilhot J, Nicolini FE, Guerci-Bresler A, Rigal-Huguet F, Maloisel F, Coiteux V, Gardembas M, Berthou C, Vekhoff A, Rea D, Jourdan E, Allard C, Delmer A, Rousselot P, Legros L, Berger M, Corm S, Etienne G, Roche-Lestienne C, Eclache V, Mahon FX, Guilhot F; SPIRIT Investigators; France Intergroupe des Leucemies Myeloides Chroniques (Fi-LMC). Imatinib plus peginterferon alfa-2a in chronic myeloid leukemia. N Engl J Med. 2010 Dec 23;363(26):2511-21. doi: 10.1056/NEJMoa1004095. PMID 21175313
- [Background] Simonsson B, Gedde-Dahl T, Markevarn B, Remes K, Stentoft J, Almqvist A, Bjoreman M, Flogegard M, Koskenvesa P, Lindblom A, Malm C, Mustjoki S, Myhr-Eriksson K, Ohm L, Rasanen A, Sinisalo M, Sjalander A, Stromberg U, Bjerrum OW, Ehrencrona H, Gruber F, Kairisto V, Olsson K, Sandin F, Nagler A, Nielsen JL, Hjorth-Hansen H, Porkka K; Nordic CML Study Group. Combination of pegylated IFN-alpha2b with imatinib increases molecular response rates in patients with low- or intermediate-risk chronic myeloid leukemia. Blood. 2011 Sep 22;118(12):3228-35. doi: 10.1182/blood-2011-02-336685. Epub 2011 Jun 17. PMID 21685374
- [Background] Hehlmann R, Lauseker M, Jung-Munkwitz S, Leitner A, Muller MC, Pletsch N, Proetel U, Haferlach C, Schlegelberger B, Balleisen L, Hanel M, Pfirrmann M, Krause SW, Nerl C, Pralle H, Gratwohl A, Hossfeld DK, Hasford J, Hochhaus A, Saussele S. Tolerability-adapted imatinib 800 mg/d versus 400 mg/d versus 400 mg/d plus interferon-alpha in newly diagnosed chronic myeloid leukemia. J Clin Oncol. 2011 Apr 20;29(12):1634-42. doi: 10.1200/JCO.2010.32.0598. Epub 2011 Mar 21. PMID 21422420
- [Background] Nicolini FE, Etienne G, Dubruille V, Roy L, Huguet F, Legros L, Giraudier S, Coiteux V, Guerci-Bresler A, Lenain P, Cony-Makhoul P, Gardembas M, Hermet E, Rousselot P, Ame S, Gagnieu MC, Pivot C, Hayette S, Maguer-Satta V, Etienne M, Dulucq S, Rea D, Mahon FX. Nilotinib and peginterferon alfa-2a for newly diagnosed chronic-phase chronic myeloid leukaemia (NiloPeg): a multicentre, non-randomised, open-label phase 2 study. Lancet Haematol. 2015 Jan;2(1):e37-46. doi: 10.1016/S2352-3026(14)00027-1. Epub 2015 Jan 7. PMID 26687426
- [Background] Burchert A, Muller MC, Kostrewa P, Erben P, Bostel T, Liebler S, Hehlmann R, Neubauer A, Hochhaus A. Sustained molecular response with interferon alfa maintenance after induction therapy with imatinib plus interferon alfa in patients with chronic myeloid leukemia. J Clin Oncol. 2010 Mar 10;28(8):1429-35. doi: 10.1200/JCO.2009.25.5075. Epub 2010 Feb 8. PMID 20142590
- [Background] Burchert A, Saussele S, Eigendorff E, Muller MC, Sohlbach K, Inselmann S, Schutz C, Metzelder SK, Ziermann J, Kostrewa P, Hoffmann J, Hehlmann R, Neubauer A, Hochhaus A. Interferon alpha 2 maintenance therapy may enable high rates of treatment discontinuation in chronic myeloid leukemia. Leukemia. 2015 Jun;29(6):1331-5. doi: 10.1038/leu.2015.45. Epub 2015 Feb 25. PMID 25712735
- [Background] Baccarani M, Rosti G, de Vivo A, Bonifazi F, Russo D, Martinelli G, Testoni N, Amabile M, Fiacchini M, Montefusco E, Saglio G, Tura S; Italian Cooperative Study Group on Myeloid Leukemia. A randomized study of interferon-alpha versus interferon-alpha and low-dose arabinosyl cytosine in chronic myeloid leukemia. Blood. 2002 Mar 1;99(5):1527-35. doi: 10.1182/blood.v99.5.1527. PMID 11861264
- [Background] Lipton JH, Khoroshko N, Golenkov A, Abdulkadyrov K, Nair K, Raghunadharao D, Brummendorf T, Yoo K, Bergstrom B; Pegasys CML Study Group. Phase II, randomized, multicenter, comparative study of peginterferon-alpha-2a (40 kD) (Pegasys) versus interferon alpha-2a (Roferon-A) in patients with treatment-naive, chronic-phase chronic myelogenous leukemia. Leuk Lymphoma. 2007 Mar;48(3):497-505. doi: 10.1080/10428190601175393. PMID 17454589
- [Background] Koskenvesa P, Kreutzman A, Rohon P, Pihlman M, Vakkila E, Rasanen A, Vapaatalo M, Remes K, Lundan T, Hjorth-Hansen H, Vakkila J, Simonsson B, Mustjoki S, Porkka K. Imatinib and pegylated IFN-alpha2b discontinuation in first-line chronic myeloid leukemia patients following a major molecular response. Eur J Haematol. 2014;92(5):413-20. doi: 10.1111/ejh.12258. Epub 2014 Jan 28. PMID 24372965
- [Background] Faderl S, Talpaz M, Estrov Z, Kantarjian HM. Chronic myelogenous leukemia: biology and therapy. Ann Intern Med. 1999 Aug 3;131(3):207-19. doi: 10.7326/0003-4819-131-3-199908030-00008. PMID 10428738
- [Background] Saussele S, Richter J, Hochhaus A, Mahon FX. The concept of treatment-free remission in chronic myeloid leukemia. Leukemia. 2016 Aug;30(8):1638-47. doi: 10.1038/leu.2016.115. Epub 2016 May 2. PMID 27133824
- [Background] Rea D, Nicolini FE, Tulliez M, Guilhot F, Guilhot J, Guerci-Bresler A, Gardembas M, Coiteux V, Guillerm G, Legros L, Etienne G, Pignon JM, Villemagne B, Escoffre-Barbe M, Ianotto JC, Charbonnier A, Johnson-Ansah H, Noel MP, Rousselot P, Mahon FX; France Intergroupe des Leucemies Myeloides Chroniques. Discontinuation of dasatinib or nilotinib in chronic myeloid leukemia: interim analysis of the STOP 2G-TKI study. Blood. 2017 Feb 16;129(7):846-854. doi: 10.1182/blood-2016-09-742205. Epub 2016 Dec 8. PMID 27932374
- [Background] Mahon, F., Richter, J., Guilhot, J., Muller, M. C., Dietz, C., Porkka, K., Hjorth-Hansen, H., Gruber, F., Panagoitidis, P., Ossenkoppele, G. J., Mayer, J., Almeida, A., Machova Polakova, K., Ehrencrona, H., Kairisto, V., Berger, M. G., Olsson stromberg, U., Mustjoki, S., Hochhaus, A., Pfirrmann, M., & Saussele, S. (2014). Interim Analysis of a Pan European Stop Tyrosine Kinase Inhibitor Trial in Chronic Myeloid Leukemia : The EURO-SKI study. Blood, 124(21), 151. Accessed March 07, 2017. Retrieved from http://www.bloodjournal.org/content/124/21/151.
- [Background] Kluin-Nelemans HC, Kester MG, van deCorput L, Boor PP, Landegent JE, van Dongen JJ, Willemze R, Falkenburg JH. Correction of abnormal T-cell receptor repertoire during interferon-alpha therapy in patients with hairy cell leukemia. Blood. 1998 Jun 1;91(11):4224-31. PMID 9596670
- [Background] Kantarjian HM, O'Brien S, Cortes JE, Shan J, Giles FJ, Rios MB, Faderl SH, Wierda WG, Ferrajoli A, Verstovsek S, Keating MJ, Freireich EJ, Talpaz M. Complete cytogenetic and molecular responses to interferon-alpha-based therapy for chronic myelogenous leukemia are associated with excellent long-term prognosis. Cancer. 2003 Feb 15;97(4):1033-41. doi: 10.1002/cncr.11223. PMID 12569603
- [Background] Hasford J, Baccarani M, Hoffmann V, Guilhot J, Saussele S, Rosti G, Guilhot F, Porkka K, Ossenkoppele G, Lindoerfer D, Simonsson B, Pfirrmann M, Hehlmann R. Predicting complete cytogenetic response and subsequent progression-free survival in 2060 patients with CML on imatinib treatment: the EUTOS score. Blood. 2011 Jul 21;118(3):686-92. doi: 10.1182/blood-2010-12-319038. Epub 2011 May 2. PMID 21536864
- [Background] Pfirrmann M, Lauseker M, Hoffmann VS, Hasford J. Prognostic scores for patients with chronic myeloid leukemia under particular consideration of competing causes of death. Ann Hematol. 2015 Apr;94 Suppl 2:S209-18. doi: 10.1007/s00277-015-2316-0. Epub 2015 Mar 27. PMID 25814087
- [Background] Rasimas J, Katsounas A, Raza H, Murphy AA, Yang J, Lempicki RA, Osinusi A, Masur H, Polis M, Kottilil S, Rosenstein D. Gene expression profiles predict emergence of psychiatric adverse events in HIV/HCV-coinfected patients on interferon-based HCV therapy. J Acquir Immune Defic Syndr. 2012 Jul 1;60(3):273-81. doi: 10.1097/QAI.0b013e31824c17c4. PMID 22728749
- [Background] Sokal JE, Cox EB, Baccarani M, Tura S, Gomez GA, Robertson JE, Tso CY, Braun TJ, Clarkson BD, Cervantes F, et al. Prognostic discrimination in "good-risk" chronic granulocytic leukemia. Blood. 1984 Apr;63(4):789-99. PMID 6584184
- [Background] Hasford J, Pfirrmann M, Hehlmann R, Allan NC, Baccarani M, Kluin-Nelemans JC, Alimena G, Steegmann JL, Ansari H. A new prognostic score for survival of patients with chronic myeloid leukemia treated with interferon alfa. Writing Committee for the Collaborative CML Prognostic Factors Project Group. J Natl Cancer Inst. 1998 Jun 3;90(11):850-8. doi: 10.1093/jnci/90.11.850. PMID 9625174
- [Background] Pfirrmann M, Baccarani M, Saussele S, Guilhot J, Cervantes F, Ossenkoppele G, Hoffmann VS, Castagnetti F, Hasford J, Hehlmann R, Simonsson B. Prognosis of long-term survival considering disease-specific death in patients with chronic myeloid leukemia. Leukemia. 2016 Jan;30(1):48-56. doi: 10.1038/leu.2015.261. Epub 2015 Sep 29. PMID 26416462
- [Background] Tateno M, Honda M, Kawamura T, Honda H, Kaneko S. Expression profiling of peripheral-blood mononuclear cells from patients with chronic hepatitis C undergoing interferon therapy. J Infect Dis. 2007 Jan 15;195(2):255-67. doi: 10.1086/509893. Epub 2006 Dec 13. PMID 17191171
- [Background] Zimmerer JM, Lesinski GB, Ruppert AS, Radmacher MD, Noble C, Kendra K, Walker MJ, Carson WE 3rd. Gene expression profiling reveals similarities between the in vitro and in vivo responses of immune effector cells to IFN-alpha. Clin Cancer Res. 2008 Sep 15;14(18):5900-6. doi: 10.1158/1078-0432.CCR-08-0846. PMID 18794103
- [Background] Osinusi A, Rasimas JJ, Bishop R, Proschan M, McLaughlin M, Murphy A, Cortez KJ, Polis MA, Masur H, Rosenstein D, Kottilil S. HIV/Hepatitis C virus-coinfected virologic responders to pegylated interferon and ribavirin therapy more frequently incur interferon-related adverse events than nonresponders do. J Acquir Immune Defic Syndr. 2010 Mar;53(3):357-63. doi: 10.1097/QAI.0b013e3181c7a29d. PMID 20101190
- [Background] Hasham A, Zhang W, Lotay V, Haggerty S, Stefan M, Concepcion E, Dieterich DT, Tomer Y. Genetic analysis of interferon induced thyroiditis (IIT): evidence for a key role for MHC and apoptosis related genes and pathways. J Autoimmun. 2013 Aug;44:61-70. doi: 10.1016/j.jaut.2013.04.002. Epub 2013 May 15. PMID 23683877
- [Background] Pfirrmann M, Hochhaus A, Lauseker M, Saussele S, Hehlmann R, Hasford J. Recommendations to meet statistical challenges arising from endpoints beyond overall survival in clinical trials on chronic myeloid leukemia. Leukemia. 2011 Sep;25(9):1433-8. doi: 10.1038/leu.2011.116. Epub 2011 May 20. PMID 21597465
- [Background] Putter H, Fiocco M, Geskus RB. Tutorial in biostatistics: competing risks and multi-state models. Stat Med. 2007 May 20;26(11):2389-430. doi: 10.1002/sim.2712. PMID 17031868